CLINICAL TRIAL: NCT00414297
Title: External Counterpulsation (ECP) for the Promotion of Collateral Growth in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: BernUniversity Hospital, Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61/06
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Artery Disease
Keywords: CAD; ECP; CFI; CPI; MPR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 ECP (Active Comparator): active ECP Therapy
  Interventions: Device: ECP Therapy
- 2 (Placebo Comparator): Sham ECP Treatment
  Interventions: Device: ECP Therapy

INTERVENTIONS:
Device: ECP Therapy — application of ECP Therapy to CAD Patients

SUMMARY:
The purpose of this study in humans with stable coronary artery disease (CAD) treatable by percutaneous coronary intervention (PCI) is to evaluate the efficacy of External Counterpulsation (ECP) with regard to the promotion of coronary collateral growth.

DETAILED DESCRIPTION:
Alternative strategies for the promotion of coronary collaterals (arteriogenesis) are a promising therapeutic alternative for at least 20% of all Patients with Coronary Artery Disease (CAD). Beside growth factors, physical exercise has been shown to improve coronary collateral function. Extracorporal Counterpulsation (ECP) mimics physical exercise in a standardized way. Before and after ECP treatment, a quantitative invasive assessment of absolute collateral flow (by calculating the CFI, i.e. Collateral Flow Index) and myocardial perfusion is performed (with calculation of the CPI, i.e. Collateral Perfusion Index and MPR, i.e. Myocardial Perfusion Reserve).

The study setting is single-blinded, sham-controlled and proceptive .

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* 1- to 3-vessel coronary artery disease (CAD)
* Stable angina pectoris
* At least 1 stenotic lesion suitable for PCI within the next 4 weeks
* No Q-wave myocardial infarction in the area undergoing CFI measurement
* Written informed consent to participate in the study

Exclusion Criteria:

* Patients admitted as emergencies
* Acute myocardial infarction within the last 3 months
* Unstable CAD
* CAD treated best by CABG
* Coronary stenotic lesion to be treated ad-hoc or within < 4 weeks
* Severe valve disease
* Pulmonary artery hypertension
* Congestive heart failure
* Atrial fibrillation
* Thrombophlebitis and/or deep vein thrombosis
* Occlusive peripheral artery disease
* Abdominal aortic aneurysm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Collateral flow index (CFI) | 21 days
Coronary collateral resistance (Rcoll) | 21 days

SECONDARY OUTCOMES:
Myocardial perfusion reserve | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof., Study Chair — University of Bern; Steffen Gloekler, MD, Principal Investigator — University of Bern
Locations (1):
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Al Kaabi A, Traupe T, Stutz M, Buchs N, Heller M. Cause or effect of arteriogenesis: compositional alterations of microparticles from CAD patients undergoing external counterpulsation therapy. PLoS One. 2012;7(10):e46822. doi: 10.1371/journal.pone.0046822. Epub 2012 Oct 8. PMID 23056467